CLINICAL TRIAL: NCT04001452
Title: 2nd International Survey on Interventional Strategies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Gabor Toth-Gayor, Principal Investigator, Medical University of Graz
Other Study IDs: ISIS 2
Record Dates: First submitted 2019-06-08; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Level of experience in interventional cardiology: Total cohort will be grouped according to experience in interventional cardiology, as defined by a single choice questionnaire:
  Yearly personal PCI volume Less than 75 / Between 75 and 150 / Between 151 and 250 / More than 250
- Level of experience with intravascular ultrasound: Total cohort will be grouped according to experience with intravascular ultrasound, as defined by a single choice questionnaire:
  General: No experience / Less than 1 year / Between 1 and 3 years / Between 3 and 5 years / More than 5 years
  Yearly: None / Less than 15 / Between 15 and 50 / More than 50
- Level of experience with optical coherence tomography: Total cohort will be grouped according to experience with optical coherence tomography, as defined by a single choice questionnaire:
  General: No experience / Less than 1 year / Between 1 and 3 years / Between 3 and 5 years / More than 5 years
  Yearly: None / Less than 15 / Between 15 and 50 / More than 50
- Level of experience with fractional flow reserve: Total cohort will be grouped according to experience with fractional flow reserve, as defined by a single choice questionnaire:
  General: No experience / Less than 1 year / Between 1 and 3 years / Between 3 and 5 years / More than 5 years
  Yearly: None / Less than 50 / Between 50 and 150 / Between 151 and 250 / More than 250
- Level of experience with non-hyperaemic pressure ratios: Total cohort will be grouped according to experience with non-hyperaemic pressure ratios, as defined by a single choice questionnaire:
  General: No experience / Less than 1 year / Between 1 and 3 years / Between 3 and 5 years / More than 5 years
  Yearly: None / Less than 50 / Between 50 and 150 / Between 151 and 250 / More than 250

SUMMARY:
The study aims to evaluate the decision-making pathways of interventional cardiologists, when assessing patients, presented with stable coronary artery disease.

DETAILED DESCRIPTION:
2nd International Survey on Interventional Strategies is a web-based platform.

The survey contains specific questions and dedicated case presentations on two major topics.

The first part queries the characteristics of the participants, including overall experience in interventional cardiology, annual volume of percutaneous coronary intervention (PCI), and duration of experience with quantitative coronary angiography (QCA), intravascular ultrasound (IVUS),optical coherence tomography (OCT), fractional flow reserve (FFR) and non-hyperaemic pressure ratios (NHPR). The survey uses here predefined categories and single-choice questions.

The second part investigates personal strategies for evaluating angiographically intermediate stenoses in the catheterization laboratory. Here, participants are asked to evaluate 5 complete coronary angiograms. All cases are characterised as stable angina without relevant changes on resting ECG. No information about non-invasive testing is known or provided.

Here participants are asked to (1) localise all relevant stenoses by indicating the involved segment; (2) define percent diameter stenosis (%DS) by visual estimate; and (3) determine the significance of the stenosis of interest. In cases of angiographic uncertainty, the preferred diagnostic tool is asked to be selected from the arsenal available in the catheterisation laboratory, namely QCA, IVUS, OCT, FFR or NHPR. Participants are asked to make their decisions assuming ideal world conditions, without considering any financial restrictions or local regulations, but only after the best clinical practice achievable in this virtual catheterisation laboratory.

ELIGIBILITY:
Inclusion criteria

* Interventional cardiologists
* Interventional cardiologists in training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be invited to join the survey via different online platforms and via social media.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Need for using any additional diagnostic tool | One month
  It will be assessed, how often participants express their desire to use one or other additional diagnostic tool to make a decision about lesion significance

SECONDARY OUTCOMES:
Need for using any additional diagnostic tool in different subgroups | One month
  It will be assessed, how often the different subgroups of participants (i.e. by age, by interventional experience, by experience with different tools) express their desire to use one or other additional diagnostic tool to make a decision about lesion significance
Accuracy of visually estimated lesion severity | One month
  Visually estimated diameter stenosis will be compared to quantitatively assessed diameter stenosis

REFERENCES:
- [Background] Toth GG, Toth B, Johnson NP, De Vroey F, Di Serafino L, Pyxaras S, Rusinaru D, Di Gioia G, Pellicano M, Barbato E, Van Mieghem C, Heyndrickx GR, De Bruyne B, Wijns W. Revascularization decisions in patients with stable angina and intermediate lesions: results of the international survey on interventional strategy. Circ Cardiovasc Interv. 2014 Dec;7(6):751-9. doi: 10.1161/CIRCINTERVENTIONS.114.001608. Epub 2014 Oct 21. PMID 25336468
- [Derived] G Toth G, Johnson NP, Wijns W, Toth B, Achim A, Fournier S, Barbato E. Revascularization decisions in patients with chronic coronary syndromes: Results of the second International Survey on Interventional Strategy (ISIS-2). Int J Cardiol. 2021 Aug 1;336:38-44. doi: 10.1016/j.ijcard.2021.05.005. Epub 2021 May 7. PMID 33971185